CLINICAL TRIAL: NCT02413944
Title: Standardized Protocol for 1µg Adrenocorticotropic Hormone (ACTH) Stimulation Test, Minimizing Technical Issues That Could Influence Test Accuracy; and Determining Salivary Free Cortisol Concentration in Healthy Controls During the Test
Brief Title: Standardized 1µg Adrenocorticotropic Hormone Stimulation Test, and Salivary Cortisol Concentration During the Test
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, leonard.saiegh, MD, Bnai Zion Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BnaiZionMC
Record Dates: First submitted 2015-02-03; First posted 2015-04-10 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- healthy volunteers (Experimental): ACTH stimulation test
  Interventions: Procedure: ACTH stimulation test

INTERVENTIONS:
Procedure: ACTH stimulation test — ACTH stimulation test

SUMMARY:
Study objectives: First, to determine whether intravenous injection of 1 mcg adrenocorticotropic hormone (ACTH) through short cannula, in healthy participants, provides reliable results of cortisol response, and whether this method would replace the conventional technique of injecting ACTH by a needle directly into a peripheral vein. Secondly, to determine salivary free cortisol concentration during the test in healthy controls.

Rationale of study: Intravenous injection of synthetic ACTH1-24 concentration through venous short cannula appears to be feasible and simple method. On the other hand, injection of ACTH1-24 by a needle directly into peripheral vein, is not infrequently complicated by technical problems in subjects with challenging veins. The investigators suppose that, both methods would have the same yield in predicting cortisol response.

Salivary free cortisol test has an evolving importance in assessing the adrenal function. This test would be reliable for use in low dose ACTH stimulation (1 mcg) test. The investigators will examine the concentration of salivary free cortisol during ACTH stimulation test, in order to determine level range in normal controls.

DETAILED DESCRIPTION:
The study will include 20 healthy participants of both sexes, aged 18-70 years, that have no clinical suspicion of hypoadrenalism, or any active medical condition or treatment that might alter blood cortisol levels. Pregnant women and patients whose medical or mental condition precludes obtaining informed consent will be excluded.

In the morning of the first visit, 1 mcg of ACTH1-24 will be injected directly into a peripheral vein. Blood and salivary samples will be drawn before injection, and 30 minutes after. Salivary cortisol will be drawn also 60 minutes after injection. At least two days later, in the morning of the second visit, 1 mcg of ACTH1-24 will be injected through short cannula in a peripheral vein, followed by injection of 5 ml of normal saline. Blood and salivary samples will be drawn before injection, and 30 minutes after. Salivary cortisol will be drawn also 60 minutes after injection. Blood cortisol results and salivary free cortisol results will be compared between tests.

ELIGIBILITY:
Inclusion Criteria:

* healthy participants of both sexes
* aged 18-70 year

Exclusion Criteria:

* any clinical suspicion of hypoadrenalism, or any active medical condition or treatment that might alter blood cortisol levels
* pregnant women and patients whose medical or mental condition precludes obtaining informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Serum cortisol concentrations during intravenous injection of 1 mcg adrenocorticotropic hormone through short cannula and during direct intravenous injection, in healthy participants. | 1 year

SECONDARY OUTCOMES:
Salivary free cortisol concentrations during intravenous injection of 1 mcg adrenocorticotropic hormone through short cannula and during direct intravenous injection, in healthy participants. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Saiegh, Principal Investigator — Bnai Zion Medical Center
Locations (1):
- Bnai Zion MC, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No